CLINICAL TRIAL: NCT05317403
Title: A Phase I Study of Venetoclax to Augment Epigenetic Modification and Chemotherapy in Pediatric and Young Adult Patients With Relapsed and Refractory Acute Myeloid Leukemia
Brief Title: Venetoclax to Augment Epigenetic Modification and Chemotherapy
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Michael Burke, Associate Professor, Department of Pediatrics, Division of Hematology/Oncology/BMT, Medical College of Wisconsin
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Venetoclax Epigenetic
Record Dates: First submitted 2022-03-08; First posted 2022-04-07 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Acute Myeloid Leukemia, in Relapse; Acute Myeloid Leukemia Refractory
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — venetoclax; Vorinostat; Cytarabine; fludarabine; Filgrastim

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- AML without Down Syndrome (Other): The subject receives 2 courses of therapy approximately 35 days each. Venetoclax: Days 1-14 Azacitidine and Vorinostat: Days 1-5 Filgrastim Days: 5 start and continue until post-nadir ANC > 500 cells/mm3 Fludarabine and Cytarabine Days 6 - 10 IT Cytarabine Day 0 or 1, optional between day 35 and 42
  Interventions: Drug: Venetoclax; Drug: Azacitadine; Drug: Vorinostat; Drug: Cytarabine; Drug: Fludarabine; Drug: Filgrastim
- AML with Down Syndrome (Other): The subject receives 2 courses of therapy approximately 35 days each. Venetoclax: Days 1-14 Azacitidine and Vorinostat: Days 1-5 Filgrastim Days: 5 start and continue until post-nadir ANC > 500 cells/mm3 Fludarabine and Cytarabine Days 6 - 10 IT Cytarabine Day 0 or 1, optional between day 35 and 42
  Interventions: Drug: Venetoclax; Drug: Azacitadine; Drug: Vorinostat; Drug: Cytarabine; Drug: Fludarabine; Drug: Filgrastim

INTERVENTIONS:
Drug: Venetoclax — Dose Level 0: Day 1 60 mg/m2 PO x1, Days 2-14 120 mg/m2/dose PO once daily (Max: 200 mg/day)
  Dose level 1: Day 1 120 mg/m2 PO x1, Days 2-14 240 mg/m2/dose PO once daily (Max: 400 mg/day)
  Dose level 2: Day 1 180 mg/m2 PO x1, Days 2-14 360 mg/m2/dose PO once daily (Max: 600 mg/day)
Drug: Azacitadine — 75 mg/m2/dose IV once daily over 15 minutes
Drug: Vorinostat — 1 year to 17.99 years old: 180 mg/m2/dose PO once daily
  ≥18 years old 200 mg PO BID. Doses should be separated by 12 hr (±4 hr)
Drug: Cytarabine — 2000 mg/m2/dose IV once daily over 3 hours
  IT Cytarabine:
  1. - 1.99 years old: 30 mg
  2. - 2.99 years old: 50 mg
     * 3 years old: 70 mg
Drug: Fludarabine — 30 mg/m2/dose IV once daily over 30 minutes
Drug: Filgrastim — 5 microgram/kg/dose subcutaneous (or IV over 15-30 min) once daily

SUMMARY:
The investigator is testing the addition of venetoclax to 5-azacitidine and vorinostat followed by standard chemotherapy to enhance treatment response in AML patients.

DETAILED DESCRIPTION:
The investigators are testing if the addition of venetoclax to epigenetic therapy will not only enhance the treatment response for patients with epigenetic lesions but improve the poor response we have observed in those patients without epigenetic lesions. The addition of venetoclax to 5-azacitidine and vorinostat followed by standard chemotherapy will be investigated. This regimen may be tolerable and increase LSC targeting resulting in deeper, more durable responses in children, adolescents, and young adults with relapsed or refractory AML

The study will enroll patients in two strata - a primary stratum of eligible patients without Down syndrome, and a secondary stratum of eligible patients with Down syndrome (DS-AML). Subjects will receive two 35 day cycles of therapy.

ELIGIBILITY:
Inclusion Criteria

* Diagnosis

  1. Patients with AML must have measurable disease (≥M1 marrow) in the bone marrow.

     * 1st or greater relapse, OR
     * Failed to go into remission after 1st or greater relapse, OR
     * Failed to go into remission from original diagnosis after 2 or more induction attempts
  2. Patients may have CNS or other sites of extramedullary disease. No cranial irradiation is allowed during the protocol therapy.
  3. Patients with treatment related AML (tAML) are eligible. A relapse of tAML is not necessary to enroll on this study thus newly diagnosed tAML are eligible.
  4. Patients with immunophenotypic AML evolving as lineage switch from ALL or acute leukemia NOS, may be eligible if they have relapsed/refractory disease
  5. Patients with Down syndrome are eligible
* Performance Level- Karnofsky > 50% for patients > 16 years of age and Lansky > 50% for patients ≤ 16 years of age. (See Appendix II for Performance Scales)
* Prior Therapy- Patients must have fully recovered from the acute toxic effects of all prior chemotherapy, immunotherapy, or radiotherapy prior to entering this study.

  1. Myelosuppressive chemotherapy
  2. Cytoreduction with hydroxyurea Hydroxyurea can be initiated and continued for up to 24 hours prior to the start of Venetoclax. It is recommended to use hydroxyurea in patients with significant leukocytosis (WBC > 50,000/L) to control blast count before initiation of systemic protocol therapy.
  3. Patients who relapsed while they are receiving cytotoxic therapy At least 7 days must have elapsed since the completion of the cytotoxic therapy, except Intrathecal chemotherapy.
  4. Hematopoietic stem cell transplant: Patients who have experienced relapse after a HSCT are eligible, provided they have no evidence of acute or chronic Graft-versus-Host Disease (GVHD), and are at least 90 days post-transplant at the time of enrollment, no longer receiving GVHD therapy.
  5. Hematopoietic growth factors: It must have been at least 7 days since the completion of therapy with GCSF or other growth factors at the time of enrollment. It must have been at least 14 days since the completion of therapy with pegfilgrastim (Neulasta®).
  6. Biologic (anti-neoplastic agent): At least 7 days after the last dose of a biologic agent. For agents that have known adverse events occurring beyond 7 days after administration, this period must be extended beyond the time during which adverse events are known to occur. The duration of this interval must be discussed with the study chair. This includes flotetuzumab.
  7. Monoclonal antibodies: At least 3 half-lives of the antibody must have elapsed after the last dose of monoclonal antibody. (i.e. Gemtuzumab = 36 days)
  8. Immunotherapy: At least 42 days after the completion of any type of immunotherapy, e.g. tumor vaccines or CAR-T cells.
  9. XRT: Craniospinal XRT is prohibited during protocol therapy. No waiting period is necessary for radiation given to non-CNS chloromas; ≥ 90 days must have elapsed if prior TBI or craniospinal XRT.
  10. Infection Prevention: Patients must be able to tolerate and receive anti-fungal prophylaxis with echinocandins or amphotericin therapy for the duration of their treatment course and neutrophil recovery (post-nadir ANC is > 750/μL).
  11. Inhibitors and Inducers ofCYP3A4

      * Patients taking strong CYP3A4 inhibitors should have their venetoclax dose reduced by 75%
      * Patients taking moderate CYP3A4 inhibitors should have their venetoclax dose reduced by 50%
      * Inhibitors of P-glycoprotein (P-gp): Patients taking p-glycoprotein inhibitors should have their venetoclax doses reduced by 50%.
* Renal and hepatic function- Patients must have adequate renal and hepatic functions as indicated by the following laboratory values:

  1. Adequate renal function defined as: Patient must have a calculated creatinine clearance or radioisotope GFR ≥ 70ml/min/1.73m2 OR a normal serum creatinine
  2. Adequate Liver Function Defined as: Direct bilirubin < 1.5 x upper limit of normal (ULN) for age or normal, AND alanine transaminase (ALT) < 5 x ULN for age. The hepatic requirements are waived for patients with known or suspected liver involvement by leukemia. This must be reviewed by and approved by the study chair or vice chair.
* Adequate Cardiac Function Defined as: Shortening fraction of ≥ 27% OR ejection fraction of ≥ 50%.
* Reproductive Function

  1. Female patients of childbearing potential must have a negative urine or serum pregnancy test confirmed within 2 weeks prior to enrollment.
  2. Female patients with infants must agree not to breastfeed their infants while on this study.
  3. Male and female patients of child-bearing potential must agree to use an effective method of contraception approved by the investigator during the study and for a minimum of 6 months after study treatment.
* Informed Consent- Patients and/or their parents or legal guardians must be capable of understanding the investigational nature, potential risks, and benefits of the study. All patients and/or their parents or legal guardians must sign a written informed consent. Age-appropriate assent will be obtained per institutional guidelines. To allow non-English speaking patients to participate in this study, bilingual health services will be provided in the appropriate language when feasible.
* Protocol Approval- All institutional, FDA, and OHRP requirements for human studies must be met.

Exclusion Criteria

•.Patients will be excluded if they have a known allergy to any of the drugs used in the study.

* Patients will be excluded if they have a systemic fungal, bacterial, viral, or other infection that is exhibiting ongoing signs/symptoms related to the infection without improvement despite appropriate antibiotics or other treatment. The patient needs to be off pressors and have negative blood cultures for 48 hours.
* Patients will be excluded if they have had any positive fungal culture within 30 days prior to enrollment or evidence of disseminated fungal disease.
* Patients will be excluded if there is a plan to administer non-protocol chemotherapy, radiation therapy, or immunotherapy during the study period.
* Patients will be excluded if they have significant concurrent disease, illness, psychiatric disorder, or social issue that would compromise patient safety or compliance with the protocol treatment or procedures, interfere with consent, study participation, follow up, or interpretation of study results.
* Patients with DNA fragility syndromes (such as Fanconi anemia, Bloom syndrome) are excluded.

Ages: 1 Year to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-03-31 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Venetoclax Dose-Limiting Toxicity | 42 months
  The primary endpoint, for dose escalation of venetoclax, is the occurrence of a dose-limiting toxicity (DLT) observed during the first course of therapy.

SECONDARY OUTCOMES:
Response Rates | 42 months
  Response rates as measured by morphologic response (CR)
Response Rates | 42 months
  Response rates as measured by morphologic response (PD)
Response Rates | 42 months
  Response rates as measured by morphologic response (SD)
Response Rates | 42 months
  Response rates as measured by morphologic response (CRi)
Response Rates | 42 months
  Response rates as measured by morphologic response (PR)
MRD | 42 months
  minimal residual disease (MRD) via multiparameter flow cytometry

CONTACTS AND LOCATIONS:
Overall Officials: Michael Burke, MD, Study Chair — Medical College of Wisconsin
Locations (1):
- Children's Wisconsin, Milwaukee, Wisconsin, United States